CLINICAL TRIAL: NCT04933747
Title: A Phase 1, Open-label, Multicenter Study to Evaluate the Pharmacokinetics of Iberdomide (CC-220) in Subjects With Renal Impairment Compared to Subjects With Normal Renal Function
Brief Title: Study to Evaluate Safety and Tolerability of Iberdomide (CC-220) in Participants With Kidney Impairment Compared to Participants With Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-CP-008
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Renal Insufficiency
Keywords: Renal Insufficiency; CC-220; Iberdomide; Phase 1
MeSH Terms: conditions — Renal Insufficiency | interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Participants with severe Renal Impairment (RI) (Experimental): Severe Renal Impairment (RI), as defined by an eGFR < 30 mL/min/1.73 m2 and not requiring dialysis, at screening
  Interventions: Drug: Iberdomide
- Group 2: Participants with kidney failure who are on intermittent hemodialysis (IHD) (Experimental): Kidney failure participants on intermittent hemodialysis (IHD)
  Interventions: Drug: Iberdomide
- Group 3: Participants with normal renal function (Experimental): Normal renal function, as defined by a creatinine clearance (Clcr) > 90 mL/min estimated using the Cockcroft-Gault (C-G) equation, at screening.
  Interventions: Drug: Iberdomide

INTERVENTIONS:
Drug: Iberdomide — Administration of a single oral dose of 1mg iberdomide in participants
  Other Names: CC-220
  Arms: Group 1: Participants with severe Renal Impairment (RI); Group 3: Participants with normal renal function
Drug: Iberdomide — Administration of a single oral dose of 1mg iberdomide in participants on 2 occasions - once on a dialysis day and once on a non-dialysis day
  Other Names: CC-220
  Arms: Group 2: Participants with kidney failure who are on intermittent hemodialysis (IHD)

SUMMARY:
This is an open-label study of iberdomide in participants with severe renal impairment or participants receiving dialysis compared to participants with normal renal function. An open-label design was selected based on the objective nature of the primary endpoints (i.e., Pharmacokinetics parameter estimates based on measurement of iberdomide and M12 concentrations). Participants with severe renal impairment (RI), participants with kidney failure on intermittent hemodialysis (IHD), and participants with normal renal function are being included in the current study. Participants with severe RI and kidney failure participants will be matched to participants with normal renal function based on sex, age (approximately ± 10 years), and body mass index (BMI; approximately ± 30%).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for All Participants (All Groups)

Participants must satisfy the following criteria to be enrolled in the study:

1. Participant is ≥ 18 and ≤ 82 years of age at the time of signing the informed consent form (ICF).
2. Participant must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Participant is able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions, the study visit schedule, and other protocol requirements, including contraception requirements.
4. Participant has a body mass index (BMI) ≥ 18 and ≤ 40 kg/m2 at screening.
5. Participant has a body weight > 50 kg at screening.
6. Participant is afebrile (febrile is defined as ≥ 38°C or 100.4°F).

   Inclusion Criteria for Participants with Severe Renal Impairment (RI) - Group 1

   Participants in Group 1 must also satisfy the following criteria to be enrolled in the study:
7. Participant has a supine systolic blood pressure (BP) ≥ 90 and ≤ 180 mm Hg, supine diastolic BP ≥ 60 and ≤ 110 mm Hg, and pulse rate ≥ 40 and ≤ 110 beats per minute.
8. Participant has severe renal impairment as defined by an eGFR < 30 mL/min/1.73 m2 (and not requiring dialysis) at screening. The eGFR will be calculated using the Modification of Diet in Renal Disease (MDRD) equation.
9. Participant must be medically stable for at least 1 month before the first IP administration with a clinically acceptable medical history, physical examination (PE), clinical laboratory safety test results, vital sign measurements, and 12-lead electrocardiograms (ECGs) consistent with the underlying stable RI condition, as judged by the Investigator.

   a. Participant must have a QTcF value < 480 ms.
10. Participant must be stable in concomitant medication regimen (defined as not starting a new medication[s] or a change in the dosage or frequency of the concomitant medication[s] within 7 days or 5 half-lives [whichever is longer] before the first IP administration).

    Inclusion Criteria for Participants with Kidney Failure on IHD - Group 2

    Participants in Group 2 must also satisfy the following criteria to be enrolled in the study:
11. Participant has a pulse rate ≥ 40 and ≤ 110 beats per minute. Blood pressure measurements must be consistent with the participant's underlying medical condition(s) and judged by the Investigator as being clinically acceptable for purposes of study entry.
12. Participant must be medically stable for at least 1 month before the first IP administration with a clinically acceptable medical history, PE, clinical laboratory safety test results, vital sign measurements, and 12-lead ECGs consistent with the underlying kidney failure, as judged by the Investigator.
13. Participant must be stable in concomitant medication regimen
14. Participant has been attending an average of 3 hemodialysis treatments per week within the 3 months prior to screening.

    Inclusion Criteria for Participants with Normal Renal Function -Group 3
15. Participant has a supine systolic BP ≥ 90 and ≤ 160 mm Hg, supine diastolic BP ≥ 50 and ≤ 100 mm Hg, and pulse rate ≥ 40 and ≤ 100 beats per minute.
16. Participant is in good health, as determined by past medical history, PE, vital signs, 12-lead ECG, and clinical laboratory safety test results, and has normal renal function, as defined by having a Clcr > 90 mL/min estimated using the C-G equation, at screening.

    1. If male, participant has a QTcF value < 470 ms;
    2. If female, participant has a QTcF value < 480 ms.
17. Participant must match at least 1 participant in Groups 1 or 2 with respect to sex, age (approximately ± 10 years), and BMI (approximately ± 30%).

Exclusion Criteria:

Exclusion Criteria for All Participants (All Groups)

The presence of any of the following will exclude a participant from enrollment:

1. Participant has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study (excluding stable renal impairment and associated comorbidities for participants in Groups 1 and 2).
2. Participant has any condition, including active or uncontrolled infection and/or the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study.
3. Participant has any condition that confounds the ability to interpret data from the study.
4. Participant has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, or excretion
5. Participant has any medical or dietary conditions affecting assessment of eGFR or creatinine clearance (not applicable for participants in Group 2).
6. Participant is a female of childbearing potential, pregnant, or breastfeeding.
7. Participant has donated blood or plasma within 8 weeks prior to the first IP administration.
8. Participant has a history of alcohol abuse within 6 months prior to the first IP administration, or positive alcohol screen.
9. Participant has history of drug abuse within 6 months prior to the first IP administration, or positive drug screen that is not consistent with the participant's prescribed medication and/or medical history.
10. Participant is known to have serum hepatitis; known to be a carrier of the hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc); - have a positive result to the test for hepatitis B or hepatitis C virus (positive viral ribonucleic acid (RNA) titer for hepatitis C) at screening or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening. Positive anti-HBc results may be further qualified with a hepatitis B virus (HBV) DNA test; subjects with non-detectable HBV levels may be included at the discretion of the Investigator.
11. Participant has been exposed to an investigational drug (new chemical entity) within 30 days prior to the first IP administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
12. Participant has consumed any medication known to be a strong CYP3A inducer (including St. John's wort) within 30 days prior to the first IP administration.
13. Participant has consumed any medication known to be a strong CYP3A inhibitor within 7 days prior to the first IP administration.
14. Participant has consumed grapefruit, grapefruit juice, or any other grapefruit-containing product or oranges, orange juice, or any other product containing and/or made from oranges within 7 days prior to the first IP administration.
15. Participant smokes more than 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
16. Participant is part of the clinical site staff personnel or a family member of the clinical site staff.
17. Participant has received immunization with a live or live attenuated vaccine within 30 days prior the first IP administration or is planning to receive immunization with a live or live attenuated vaccine within 30 days following administration of the last dose of IP.
18. Participant has a history of multiple drug allergies or drug-related anaphylaxis.

    Exclusion Criteria for Participants with Severe Renal Impairment and Participants with Kidney Failure on IHD - Groups 1 and 2

    The presence of any of the following will also exclude a participant from enrollment:
19. Participant has any serious and/or unstable medical condition occurring within 3 months prior to screening (excluding stable renal impairment and associated comorbidities) with complete resolution of any symptoms and no sequelae that would place the participant at a higher risk from receiving IP, based on Investigator assessment in consultation with the Medical Monitor.
20. Participant has any clinically significant laboratory abnormality not related to renal impairment and related complications.
21. Participant has a history of renal transplant.

    a. Participants who had a renal transplant approximately > 2 years which is no longer functioning are allowable.

    Exclusion Criteria for Participants with Normal Renal Function - Group 3

    The presence of any of the following will also exclude a participant from enrollment:
22. Participant has used any prescribed systemic or topical medication within 30 days prior to the first dose administration.
23. Participant has used any non-prescribed systemic or topical medication within 14 days prior to the first dose administration.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Iberdomide Pharmacokinetics - AUC(0-T) | Up to 72 hours following the last dose of iberdomide
  Estimation of area under the plasma concentration -time curve (AUC) calculated from time zero to time t, where t is the time point of the last measurable concentration
Metabolite M12 Pharmacokinetics - AUC(0-T) | Up to 72 hours following the last dose of iberdomide
  Estimation of AUC calculated from time zero to time t, where t is the time point of the last measurable concentration
Iberdomide Pharmacokinetics - AUC(INF) | Up to 72 hours following the last dose of iberdomide
  Estimation of AUC calculated from time zero extrapolated to infinity
Metabolite M12 Pharmacokinetics - AUC(INF) | Up to 72 hours following the last dose of iberdomide
  Estimation of AUC calculated from time zero extrapolated to infinity
Iberdomide Pharmacokinetics - Cmax | Up to 72 hours following the last dose of iberdomide
  Estimation of maximum observed plasma concentration
Iberdomide Pharmacokinetics - Tmax | Up to 72 hours following the last dose of iberdomide
  Estimated time to Cmax
Metabolite M12 Pharmacokinetics - Tmax | Up to 72 hours following the last dose of iberdomide
  Estimated time to Cmax
Iberdomide Pharmacokinetics - T-HALF | Up to 72 hours following the last dose of iberdomide
  Estimation of terminal elimination half-life in plasma
Metabolite M12 Pharmacokinetics - T-HALF | Up to 72 hours following the last dose of iberdomide
  Estimation of terminal elimination half-life in plasma
Iberdomide Pharmacokinetics - CLT/F | Up to 72 hours following the last dose of iberdomide
  Apparent total plasma clearance when dosed orally
Iberdomide Pharmacokinetics - CLNR/F | Up to 72 hours following the last dose of iberdomide
  Apparent nonrenal clearance
Iberdomide Pharmacokinetics - VZ/F | Up to 72 hours following the last dose of iberdomide
  Estimation of apparent volume of distribution when dosed orally
Iberdomide Pharmacokinetics - CLR | Up to 72 hours following the last dose of iberdomide
  Renal Clearance
Metabolite M12 Pharmacokinetics - CLR | Up to 72 hours following the last dose of iberdomide
  Renal clearance
Iberdomide Pharmacokinetics - UR | Up to 72 hours following the last dose of iberdomide
  Estimation of amount excreted in urine
Iberdomide Pharmacokinetics - CLD | 4 hours post-start of dialysis
  Dialysis clearance

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | From enrollment until at least 28 days after completion of the study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values), regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution - 001, Orlando, Florida
  - Local Institution - 002, Knoxville, Tennessee
  - Local Institution - 003, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm